CLINICAL TRIAL: NCT03143712
Title: An Open Label Study to Compare the Oral Bioavailability of a Tablet of GLPG1690 Relative to a Capsule After Single-dose Intake in Healthy Subjects and to Evaluate the Effect of Food on the Tablet
Brief Title: Study to Assess Bioavailability of GLPG1690 Given as Oral Capsule or Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1690-CL-103
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG1690

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): GLPG1690 oral capsules after breakfast
  Interventions: Drug: GLPG1690
- Treatment B (Experimental): GLPG1690 oral tablets after breakfast
  Interventions: Drug: GLPG1690
- Treatment C (Experimental): GLPG1690 oral tablets after overnight fast
  Interventions: Drug: GLPG1690

INTERVENTIONS:
Drug: GLPG1690 — Oral administration of GLPG1690 in three different treatment conditions (treatment A through C)

SUMMARY:
This study is a Phase I, randomized, open-label, cross-over study with three single-dose treatments to compare the bioavailability of an oral tablet relative to an oral capsule of GLPG1690 after single dose intake in healthy male subjects and to evaluate the effect of food on the bioavailability of the oral tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18-50 years of age, inclusive
2. Body mass index (BMI) between 18-30 kg/m2, inclusive, with a weight of at least 50 kg.
3. Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and laboratory findings.
4. Discontinuation of all medications except occasional paracetamol at least 2 weeks or 5 half-lives prior to the first study drug administration
5. Non-smokers and not using any nicotine-containing products.
6. Negative urine drug screen and alcohol breath test.
7. Current sexually active male agrees to use adequate contraception/preventive exposure measures from the time of first dose of study drug, during the study and until 12 weeks after the last study drug dose.
8. Subjects should be willing to consume the non-vegetarian high-fat and high-calorie breakfast.
9. Able and willing to sign the ICF

Exclusion Criteria:

1. Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug
2. Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or any history of hepatitis from any cause with the exception of hepatitis A.
3. History of or a current immunosuppressive condition.
4. Presence of abnormal liver function. Diagnosis of disease of Gilbert is accepted. Retesting is allowed.
5. Renal function with an estimated creatinine clearance <80 ml/min based on the Cockcroft-Gault formula. Retesting is allowed.
6. Presence of any condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
7. History of malignancy within the past 5 years
8. Clinically relevant abnormalities detected on ECG regarding either rhythm or conduction (e.g., QTcF >450 ms, or a known long QT syndrome).
9. Clinically relevant abnormalities detected on vital signs.
10. Dietary requirements precluding participation in the study
11. Significant blood loss (including blood donation [≥450 mL]), or transfusion of any blood product within 8 weeks prior to the signing of ICF.
12. Active drug or alcohol abuse within 2 years prior to the initial study drug administration.
13. Consumption of large quantities of caffeinated coffee or tea (>6 cups/day), or equivalent.
14. Concurrent participation or participation in a drug or drug/device investigational research study.
15. Subjects who participated in a previous study with the same compound (GLPG1690).
16. Investigator or any sub-investigator, or other staff or relative.
17. Any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Assessment of the maximum observed plasma concentration of GLPG1690 after single oral doses | predose at day 1 and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours post dosing
  Determine the bioavailability of GLPG1690 by assessing PK parameters
Assessment of the time to reach the maximum observed plasma concentration of GLPG1690 after single oral doses | predose at day 1 and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours post dosing
  Determine the bioavialability of GLPG1690 by assessing PK parameters
Assessment of the time of the last quantifiable plasma concentration of GLPG1690 after single oral doses | predose at day 1 and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 and 48 hours post dosing
  Determine the bioavialability of GLPG1690 by assessing PK parameters

SECONDARY OUTCOMES:
The number of subjects with adverse events | Throughout the study from screening until the follow up visit (day 7 of dosing period 3)
  To assess safety and tolerability of GLPG1690
The number of subjects with abnormal vital signs | Throughout the study from screening until the follow up visit (day 7 of dosing period 3)
  To assess safety and tolerability of GLPG1690
The number of subjects with abnormal ECG | Throughout the study from screening until the follow up visit (day 7 of dosing period 3)
  To assess safety and tolerability of GLPG1690
The number of subjects with abnormal physical examination | Throughout the study from screening until the follow up visit (day 7 of dosing period 3)
  To assess safety and tolerability of GLPG1690
The number of subjects with abnormal laboratory analysis | Throughout the study from screening until the follow up visit (day 7 of dosing period 3)
  To assess safety and tolerability of GLPG1690

CONTACTS AND LOCATIONS:
Overall Officials: Ann Fieuw, MD MSc, Study Director — Galapagos NV
Locations (1):
- SGS CPU, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Aar E, Desrivot J, Dupont S, Heckmann B, Fieuw A, Stutvoet S, Fagard L, Van de Wal K, Helmer E. Safety, Pharmacokinetics, and Pharmacodynamics of the Autotaxin Inhibitor GLPG1690 in Healthy Subjects: Phase 1 Randomized Trials. J Clin Pharmacol. 2019 Oct;59(10):1366-1378. doi: 10.1002/jcph.1424. Epub 2019 Apr 23. PMID 31012984